CLINICAL TRIAL: NCT01636414
Title: Reinfusion Drains vs Tranexamic Acid in Total Joint Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 051114B; NCT01514474 (obsolete NCT alias)
Record Dates: First submitted 2012-06-14; First posted 2012-07-10 (Estimated); Results first posted 2016-04-25 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-07

CONDITIONS: Total Joint Arthroplasty
Keywords: Total joint arthroplasty, blood loss
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hemovac drain (Active Comparator)
  Interventions: Procedure: Hemovac drain
- Re-infusion drain (Active Comparator)
  Interventions: Procedure: Re-infusion drain
- Tranexamic drain (Active Comparator)
  Interventions: Procedure: Tranexamic drain

INTERVENTIONS:
Procedure: Hemovac drain — The Hemovac drain is a device placed under your skin used to collect blood during surgery.
  Arms: Hemovac drain
Procedure: Re-infusion drain — This device is used during and after surgery to collect blood lost during this time and prepares the blood for possible reinfusion.
  Arms: Re-infusion drain
Procedure: Tranexamic drain — Tranexamic Acid is a synthetic amino acid that prevents the breakdown of blood clots which reduces bleeding.
  Arms: Tranexamic drain

SUMMARY:
It is widely reported that a large percentage of total joint replacement patients receive allogeneic (human donor blood) blood transfusions due to perioperative blood loss with numbers ranging from 30% to 80%.

The risks of allogenic blood transfusion are well documented in the literature. In addition, they are time-consuming: often lengthening hospital stay and decreasing the availability for postoperative physical therapy. Moreover, they are costly at several hundred dollars per unit, and allogeneic transfusions are linked with immunosuppression and increased postoperative infection rates and wound healing problems, which are devastating complications in this elective, joint replacement population. Several options are available for diminishing the need for allogenic blood transfusion following elective total joint replacement. These include the use of perioperative blood salvage devices (OrthoPAT) and tranexamic acid. While there is data to support the use of both OrthoPat and Tranexamic acid in primary total joint arthroplasty, there is little information comparing one versus the other in terms of efficacy and economics.

The purpose of this study is to compare the safety, effectiveness and cost benefit of Hemovac drain, OrthoPAT and Tranexamic Acid to manage blood loss during total hip and total knee replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting for primary unilateral hip or knee arthroplasty
2. > 18 years of age
3. Preoperative hemoglobin on day of surgery > 10mg/dL

Exclusion Criteria:

1. Patients with a preoperative Hgb < 10mg/dL
2. Patients who are unwilling to consent to blood transfusions
3. Patients with a history of bleeding disorder
4. Patients on anticoagulation therapy preoperatively (ASA 325mg, Plavix or Coumadin)
5. Patients with a history of Thromboembolic events ( DVT, PE, CVA MI)
6. Patients with platelet counts < 100,000
7. Patients with kidney disease (Serum Cr > 1.2)
8. Patients with end stage renal disease or on hemodialysis
9. Patients with renal transplant
10. Patients presenting for bilateral total hip or knee arthroplasty
11. Patients presenting for conversion or revision total hip or knee procedures
12. Patients donating pre-autologous blood
13. Patients with primary hematologic disease or malignancy
14. Patients with allergy to Tranexamic Acid
15. Patients with hepatic disease
16. Patients not discontinuing steroid use prior to surgery
17. Patients with religious beliefs/practices prohibiting blood transfusions
18. Patients with cognitive impairment
19. Patients who are terminally ill

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2012-05; Primary Completion 2014-06 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- OrthoCarolina, PA, Charlotte, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hemovac Drain | Re-infusion Drain | Tranexamic Drain
Started | 64 | 66 | 74
Completed | 61 | 60 | 65
Not Completed | 3 | 6 | 9

BASELINE CHARACTERISTICS:
Population: All patients who completed the study are included in the reported results. Patients that were withdrawn from the study did not receive treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hemovac Drain | Re-infusion Drain | Tranexamic Drain | Total
Number analyzed (Participants) | 61 | 60 | 65 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.03 (8.21) | 63.77 (7.87) | 61.07 (14.31) | 62.68 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 43 | 38 | 106
  Male | 36 | 17 | 27 | 80

OUTCOME MEASURES:

1. Primary Outcome: Blood Transfusion
Description: Transfusion Rate (i.e, number of participants needing Blood Transfusion) Between Treatment Groups
Time Frame: Inpatient Postoperative, on average 3 days after surgery
Measure: Number; unit: participants
Arm/Group | Hemovac Drain | Re-infusion Drain | Tranexamic Drain
Number analyzed (Participants) | 61 | 60 | 65
participants | 5 | 8 | 1

2. Primary Outcome: Change in Hemoglobin Level
Description: Change in hemoglobin following surgery. Initial (baseline) measure was prior to surgery on day of surgery. Follow-up measurement occurred the day following surgery.
Time Frame: Post-operative on day 2 (first day after surgery)
Measure: Median (Inter-Quartile Range); unit: g/dl
Arm/Group | Hemovac Drain | Re-infusion Drain | Tranexamic Drain
Number analyzed (Participants) | 61 | 60 | 65
g/dl | -3.95 [-5.0 to -3.1] | -3.80 [-4.7 to -3.1] | -2.90 [-3.80 to -2.0]

ADVERSE EVENTS:
Arm/Group | Hemovac Drain | Re-infusion Drain | Tranexamic Drain
Serious Adverse Events (participants affected / at risk) | 1/61 | 0/60 | 1/65
Other Adverse Events (participants affected / at risk) | 2/61 | 0/60 | 1/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hemovac Drain (N=61) | Re-infusion Drain (N=60) | Tranexamic Drain (N=65)
Occluded superficial femoral artery (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Reoperation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) — Reoperation during index hospitalization stay
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hemovac Drain (N=61) | Re-infusion Drain (N=60) | Tranexamic Drain (N=65)
Extended hospitalization (Surgical and medical procedures) | 2 (2) | 0 | 1 (1) — Extended hospitalization stay, beyond the standard of care of 3 post-operative days.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No